CLINICAL TRIAL: NCT00711126
Title: A Single-centre, Open-label, Sequential, Dose-ascending Study to Examine Safety, Tolerability, Pharmacodynamics and Pharmacokinetics of Single Intravenous, Inhaled and Oral Doses of GW642444 in Healthy Male Subjects
Brief Title: A Study To Investigate Safety, Blood Levels And Effects Of Giving GW642444, By Mouth, By Inhalation & By Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2C106180
Record Dates: First submitted 2008-07-03; First posted 2008-07-08 (Estimated); Last update posted 2017-07-21 (Actual); Status verified 2017-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: intravenous,; tolerability; pharmacokinetics,; oral,; pharmacodynamics,; safety,; GW642444,; inhaled,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Arm 1 (Experimental): HVTs
  Interventions: Drug: GW642444
- Arm 2 (Experimental): HVTs
  Interventions: Drug: GW642444
- Arm 3 (Experimental): HVTs
  Interventions: Drug: GW642444
- Arm 4 (Experimental): HVTs
  Interventions: Drug: GW642444
- Arm 5 (Experimental): HVTs
  Interventions: Drug: GW642444
- Arm 6 (Experimental): HVTs
  Interventions: Drug: GW642444

INTERVENTIONS:
Drug: GW642444 — 2.5mcg IV
  Arms: Arm 1
Drug: GW642444 — 5mcg IV
  Arms: Arm 2
Drug: GW642444 — 10mcg IV
  Arms: Arm 3
Drug: GW642444 — 100mcg inhaled
  Arms: Arm 4
Drug: GW642444 — 20mcg IV
  Arms: Arm 5
Drug: GW642444 — 500mcg oral
  Arms: Arm 6

SUMMARY:
This study will involve the use of a new medicine called GW642444 being developed for the treatment of asthma and chronic obstructive pulmonary disease (COPD). The purpose of the study is to see how safe and how well tolerated the study drug is when it is given as a liquid by mouth or by injection into a vein. In addition the study will measure how much of the medicine gets into the bloodstream when it is given by mouth, by injection into a vein and inhaled, and how long the body takes to get rid of it.

DETAILED DESCRIPTION:
This will be a single-centre, open-label, dose-ascending study in 9 healthy male subjects to establish safe and well tolerated systemic exposure safety margins for GW642444 following intravenous and oral dosing to support future studies. Additionally a single inhaled dose of GW642444M will be administered to provide data to estimate inhaled bioavailability of GW642444 and the extent of renal excretion following dosing via this route. It is planned to administer four, dose-ascending, intravenous administrations of GW642444 during treatment periods 1, 2, 3 and 5; the inhaled dose would be administered in treatment period 4 and the oral dose in treatment period 6. The sequence of treatment administration may be altered if required for logistical reasons, however doses of intravenous and oral GW642444 will be administered strictly in dose ascending order. All intravenous doses will be administered as an infusion given at a constant rate over a 1 hour period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with laboratory parameters outside the reference range for this age group may be included only if the Investigator considers the finding will not introduce risk factors and will not interfere with the study procedures.
* Male between 18 and 65 years of age.
* Body weight ≥ 50 kg and Body Mass Index (BMI) within the range 19 - 29.9 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* No significant abnormality on 12-lead electrocardiogram (ECG) at screening
* Demonstrated ability to use the inhaler device in a satisfactory and repeatable manner.
* Subjects who are current non-smokers who have not used any tobacco products in the 6-month period preceding the screening visit and have a pack history of ≤ 10 pack years.

Exclusion Criteria:

* Any clinically relevant abnormality identified at the screening medical assessment (physical examination/medical history), clinical laboratory tests, or ECG.
* A screening Holter ECG tracing that reveals clinically concerning arrhythmias.
* A history of elevated supine blood pressure or a mean supine blood pressure persistently equal to or higher than 140/90 mmHg at screening.
* A mean heart rate outside the range 45- 90 beats per minute (bpm) at screening.
* Where participation in the study would result in donation of blood in excess of 500 millilitres (mL) within a 3 month period.
* The subject has participated in a clinical study with a New Chemical Entity (NCE), or any other drug within a clinical study, within the past 3 months.
* The subject has a history of drug or other allergy, which, in the opinion of the responsible physician, contraindicates their participation.
* Any adverse reaction including immediate or delayed hypersensitivity to any β2 (beta) agonist or sympathomimetic drug, or known or suspected sensitivity to the constituents of GW642444 inhalation powder (for example; lactose, magnesium stearate).
* The subject has a positive pre-study drug/alcohol screen. A minimum list of drugs that will be screened for include amphetamines, barbiturates, cocaine, opiates, cannabinoids and benzodiazepines.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening (with the exception of phase I hepatic impairment studies, oncology studies, hepatitis, hepatic fibrosis, or Human Immunodeficiency Virus (HIV) studies).
* A positive test for HIV antibody.
* History of regular alcohol consumption within 6 months of the study defined as:
* an average weekly intake of greater than 21 units or an average daily intake of greater than 3 units. One unit is equivalent to a half-pint (220mL) of beer or 1 (25mL) measure of spirits or 1 glass (125mL) of wine.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Unwillingness or inability to follow the procedures outlined in the protocol.
* Urinary cotinine levels (or Carbon Monoxide (CO) breath monitoring) indicative of smoking or history or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and/or pommelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-10-21 (Actual); Primary Completion 2008-12-17 (Actual); Study Completion 2008-12-17 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of GW642444M (key assessments include: measurements of heart rate, blood pressure, electrocardiogram (ECG) (including QTc assessments), lead II monitoring, potassium and glucose, laboratory safety data and review of adverse events | Various

SECONDARY OUTCOMES:
Plasma PK parameters for IV, inhaled and oral routes of administration | Various
Urine PK parameters for the intravenous and inhaled routes of administration | Various

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Harrell AW, Siederer SK, Bal J, Patel NH, Young GC, Felgate CC, Pearce SJ, Roberts AD, Beaumont C, Emmons AJ, Pereira AI, Kempsford RD. Metabolism and disposition of vilanterol, a long-acting beta(2)-adrenoceptor agonist for inhalation use in humans. Drug Metab Dispos. 2013 Jan;41(1):89-100. doi: 10.1124/dmd.112.048603. Epub 2012 Oct 4. PMID 23043183
- See also: Results for study B2C106180 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/B2C106180?search=study&search_terms=B2C106180#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Individual Participant Data Set: B2C106180 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: B2C106180 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: B2C106180 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: B2C106180 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: B2C106180 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: B2C106180 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: B2C106180 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register